CLINICAL TRIAL: NCT05963945
Title: Multi-Reader Retrospective Study Examining Carebot AI CXR 2.0.21-v2.01 Implementation in Everyday Radiology Clinical Practice
Status: Completed | Type: Observational
Sponsor: Carebot s.r.o. (Industry)
Responsible Party: Sponsor
Other Study IDs: 00002
Record Dates: First submitted 2023-07-12; First posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Pneumothorax; Pulmonary Nodule, Solitary; Atelectasis; Subcutaneous Emphysema; Cardiomegaly; Consolidation; Pleural Effusion
Keywords: Artificial Intelligence; Computer-Aided Detection; Deep Learning; Chest X-ray; Radiology
MeSH Terms: conditions — Pneumothorax; Solitary Pulmonary Nodule; Pulmonary Atelectasis; Subcutaneous Emphysema; Cardiomegaly; Pleural Effusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective collection for the period October 18th, 2022, and November 17th, 2022: A total of 1,073 chest X-rays were acquired within the specified period at the department. The data collection remained intact and unaffected throughout the testing phase, ensuring the integrity of the dataset. The collected sample accurately represents the prevalence of findings within the observed population. After excluding ineligible studies such as X-rays from patients under 18 years of age, lateral projection X-rays, and scans of insufficient quality, a total of 956 relevant CXRs were identified for further assessment.
  Interventions: Device: Carebot AI CXR

INTERVENTIONS:
Device: Carebot AI CXR — The proposed DLAD (Carebot AI CXR) is a deep learning-based medical device designed to assist radiologists in interpreting chest X-ray images acquired in anteroposterior (AP) or posteroanterior (PA) projection. By employing advanced deep learning algorithms, this solution enables automatic detection of abnormal findings by analyzing visual patterns associated with specific conditions. The targeted abnormalities include atelectasis (ATE), consolidation (CON), pleural effusion (EFF), pulmonary lesion (LES), subcutaneous emphysema (SCE), cardiomegaly (CMG), and pneumothorax (PNO). The DLAD functions as a prediction algorithm complemented by various application peripherals, such as web-based communication tools, DICOM file conversion capabilities, and storage and reporting libraries supporting both DICOM Structured Report and DICOM Presentation State formats.

SUMMARY:
The primary objective is to evaluate the performance parameters of the proposed DLAD (Carebot AI CXR) in comparison to individual radiologists.

DETAILED DESCRIPTION:
In the period between October 18th, 2022, and November 17th, 2022, anonymized chest X-ray images of patients were collected at the Radiodiagnostic Department of the Havířov Hospital, p.o. The collection process involved utilizing the CloudPACS imaging and archiving system provided by OR-CZ spol. s r.o.

The collected X-ray images were subjected to the proposed DLAD (Carebot AI CXR) for analysis. Subsequently, the DLAD's performance was compared with the standard clinical practice, where radiologists assessed the CXR images in the simulated hospital setting with access to standard viewing tools (e.g., pan, zoom, WW/WL) and were given an unlimited amount of time to complete the review. Each radiologist determined the presence or absence of 7 indicated radiological findings, including atelectasis (ATE), consolidation (CON), pleural effusion (EFF), pulmonary lesion (LES), subcutaneous emphysema (SCE), cardiomegaly (CMG), and pneumothorax (PNO).

ELIGIBILITY:
Inclusion Criteria:

* Hospital patients > 18 years who were referred for chest radiography October 18th, 2022, and November 17th, 2022 at the Radiodiagnostic Department of the Havířov Hospital, p.o.

Exclusion Criteria:

* Patients < 18 years
* Chest X-ray images in lateral positions
* Duplicated chest X-ray images

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient's Sex Female: 480 (50.21 %) Male: 474 (49.58 %) Unspecified: 2 (0.21 %)
  Patient's Age 18-30: 58 (6.07 %) 31-50: 163 (17.05 %) 51-70: 366 38.28 %) 70+: 369 (38.60 %)
Sampling Method: Non-Probability Sample
Enrollment: 956 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2022-11-17 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Performance test | March 2023
  The primary objective is to evaluate the performance parameters of the proposed DLAD (Carebot AI CXR) in comparison to individual radiologists. The performance test includes sensitivity and specificity, positive and negative likelihood ratio, and positive and negative predictive value. The aforementioned parameters are statistically compared using confidence intervals (CI) and p-Values. The comparison procedure consists of two steps: a global hypothesis test is conducted to determine whether there are significant differences between DLAD and radiologists. If the global hypothesis test yields a significant result, individual hypothesis tests are performed. Additionally, multiple comparison methods, such as McNemar with continuity correction for Se and Sp, Holm method for LRs, and weighted generalized score statistics for PVs, are applied to control the overall error rate. All tests are performed as two-tailed tests at the 5% significance level.

CONTACTS AND LOCATIONS:
Locations (1):
- Nemocnice Havířov, p. o., Havířov, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] KVAK, Daniel, Anna CHROMCOVÁ, Petra OVESNÁ, Jakub DANDÁR, Marek BIROŠ, Robert HRUBÝ, Daniel DUFEK a Marija PAJDAKOVIĆ. Can Deep Learning Reliably Recognize Abnormality Patterns on Chest X-rays? A Multi-Reader Study Examining One Month of AI Implementation in Everyday Radiology Clinical Practice. arXiv. 2023, 2305.10116, 26 s.